CLINICAL TRIAL: NCT01398332
Title: Global Registry for Endovascular Aortic Treatment (GREAT)
Brief Title: Evaluation of the GORE® C3 Delivery System Module
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: GRT 10-12
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Aortic pathologies: Indication for aortic endovascular stent graft repair
  Interventions: Device: Stent graft (EXCLUDER)

INTERVENTIONS:
Device: Stent graft (EXCLUDER) — Endovascular repair
  Other Names: EXCLUDER

SUMMARY:
This is an observational Registry designed to obtain early data on the use of the GORE® EXCLUDER® AAA Endoprosthesis with C3 Delivery System.

DETAILED DESCRIPTION:
This is a retrospective and prospective observational cohort Registry designed to obtain data on the use of the GORE® EXCLUDER® AAA Endoprosthesis with C3 Delivery System. Patient and device performance outcomes will be collected during treatment and throughout all post-treatment visits, including follow-up extending up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age required by local regulations (as applicable)
2. Indication for aortic endovascular stent graft repair as determined by the treating physician (refer to current Instructions for Use of the GORE® EXCLUDER® AAA Endoprosthesis with C3 Delivery System)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergo endovascular treatment for aortic pathologies with the GORE® EXCLUDER® AAA Endoprosthesis with C3 Delivery System.
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2011-01; Primary Completion 2024-07 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Evaluate procedural outcomes for the GORE® EXCLUDER® AAA Endoprosthesis with C3 Delivery System when used in accordance with the standard medical practice at each participating hospital. | Up to 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Verhoeven, MD, Principal Investigator — Klinikum Nürnberg-Süd
Locations (1):
- Klinikum Nürnberg-Süd, Nuremberg, Germany